CLINICAL TRIAL: NCT00060957
Title: Botulinum Toxin for Spasticity in Cerebral Palsy
Brief Title: Botulinum Toxin (BOTOX) for Cerebral Palsy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1R01HD035750-01 (NIH)
Record Dates: First submitted 2003-05-16; First posted 2003-05-19 (Estimated); Last update posted 2016-09-26 (Estimated); Status verified 2011-05

CONDITIONS: Cerebral Palsy; Muscle Spasticity
Keywords: Cerebral Palsy; Spasticity; Botulinum toxin; BOTOX
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity | interventions — Botulinum Toxins, Type A

INTERVENTIONS:
Drug: Botulinum toxin type A

SUMMARY:
This study examines botulinum toxin (BOTOX, or BTX) for the treatment of muscle twitches and spasticity associated with cerebral palsy in children. Botulinum toxin is a naturally occurring bacterial toxin (botulinum toxin) that inactivates certain parts of muscles.

DETAILED DESCRIPTION:
This trial will test the effectiveness of BTX injections versus placebo to reduce plantar-flexor spasticity and improve function and mobility in children with spastic diplegia, a common form of cerebral palsy. The study will evaluate the effects of the treatment across five domains that relate to disability: pathophysiology, impairment, functional limitation, disability, and societal limitation.

Forty children, ages 4 to 12 years, will be recruited and randomized into one of two groups. Group A will receive BTX. Group B will receive a placebo injection. Participants will be assessed at the beginning of the trial and at Weeks 3, 8, 12, and 24. Assessments include quantitative electromyographic kinesiology measurements, electromechanical measurement of joint torque across the ankle joint using the Spasticity Measurement System, Gross Motor Function Measure, physical exam parameters, energy expenditure using the Energy Cost Index, kinematic gait analysis, and the Canadian Occupational Performance Measure.

Participants are followed for a total of 6 months. Participants initially randomized to Group B will have the opportunity for BTX treatment after 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Spastic diplegic cerebral palsy
* Community or independent ambulators
* Expressive communication skills at age 3 or above
* Stable social environment
* Reasonable proximity to the medical center
* Physical therapy at least once per week
* No other serious health problems that would interfere with the study

Exclusion Criteria:

* Other forms of cerebral palsy
* Previous treatment with botulinum toxin
* Musculoskeletal contractures greater than 15 degrees
* Unstable social environment

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40
Dates: Start 1997-07; Primary Completion 2002-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ross M. Hays, M.D., Principal Investigator — Children's Hospital and Regional Medical Center
Locations (1):
- Children's Hospital and Regional Medical Center, Seattle, Washington, United States